CLINICAL TRIAL: NCT04948476
Title: Promoting Kidney Recovery After Acute Kidney Injury Receiving Dialysis
Acronym: Recover-AKI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samuel Silver (Other)
Collaborators: Unity Health Toronto (Other)
Responsible Party: Sponsor-Investigator, Samuel Silver, Dr. Samuel A Silver, Queen's University
Organization: Queen's University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6027699
Record Dates: First submitted 2021-06-24; First posted 2021-07-02 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standardized Dialysis and Structured Discontinuation (S2D2) (Experimental): Prescription to minimize dialysis-induced ischemia and standardize dialysis discontinuation
  Interventions: Other: Standardized Dialysis and Structured Discontinuation (S2D2)
- Usual Care (Active Comparator): Dialysis prescription ordered by their primary nephrologist/intensivist.
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Standardized Dialysis and Structured Discontinuation (S2D2) — Prescription to minimize dialysis-induced ischemia
  * Cool dialysate (35.0◦C)
  * Dialysate sodium of 145mmol/L
  * Dialysate calcium of 1.5mmol/L
  * Maximum ultrafiltration rate of 10mL/kg/hour (if no weight, maximum is 500mL/hour)
    * Note: If dialysis machines cannot get to the specified values, values closest to these are acceptable.
  Structured dialysis discontinuation (all criteria met)
  * Most recent pre-dialysis potassium <6mmo/L and bicarbonate >12mmol/L
  * Most recent urine volume ≥1L/day OR last ultrafiltration on dialysis <1L/session
  * If available, timed urine collection with result for mean creatinine and/or urea clearance >12mL/min
  Arms: Standardized Dialysis and Structured Discontinuation (S2D2)
Other: Usual Care — Dialysis prescription ordered by their clinical team. Decisions on dialysis discontinuation will be left to individual clinicians and will not be guided by a standard protocol.
  Arms: Usual Care

SUMMARY:
The overall goal of this study is to evaluate the feasibility of conducting a randomized controlled trial comparing a standardized dialysis strategy versus usual care (dialysis prescription ordered by each patient's primary nephrologist) in patients with AKI-receiving dialysis.

ELIGIBILITY:
Inclusion Criteria:

* Received ≥2 sessions of any dialysis modality for presumed AKI
* Plans for continued intermittent hemodialysis or sustained low efficiency dialysis treatments

Exclusion Criteria:

1. Receipt of dialysis for ≥90 days
2. Known baseline estimated glomerular filtration rate (eGFR) <15mL/min/1.73m2
3. Strong clinical suspicion of urinary tract obstruction, rapidly progressive glomerulonephritis (RPGN), vasculitis, thrombotic microangiopathy (TMA), myeloma related cast nephropathy, or acute interstitial nephritis (AIN) as the underlying cause of AKI
4. Receipt of any dialysis prior to the current admission within the past 2 months
5. Kidney transplant within the past 12 months
6. Pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2022-04-12 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
Recruitment | 2 years
  Recruitment of the target population to the RCT
Fidelity | 2 years
  At least 80% of randomized participants remain in the trial and on the allocated study treatment

SECONDARY OUTCOMES:
Dialysis-Free Days | 6-months
  The number of days that a patient did not need dialysis. A patient can only accrue dialysis-free days after the final dialysis session that commences the monitoring period for kidney recovery. Participants who die will be considered to have zero dialysis-free days.
Hypotensive Event on Dialysis | 6-months
  Defined as a drop in blood pressure requiring one of:
  * Initiation of a vasopressor during renal replacement therapy (RRT) session, OR,
  * Premature discontinuation of RRT session due to blood pressure drop, OR,
  * Any other intervention to stabilize blood pressure during the dialysis session as noted in the nursing record

OTHER OUTCOMES:
Arrhythmia on Dialysis | 6-months
  Defined as new atrial (excluding sinus tachycardia or sinus arrhythmia) or ventricular arrhythmia that develops during RRT and was not present prior to the initiation of RRT

CONTACTS AND LOCATIONS:
Overall Officials: Samuel A Silver, Principal Investigator — Queen's University
Locations (1):
- Kingston Health Sciences Centre, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Deidentified patient data will be available up to 3 years after manuscript publication to researchers with methodologically sound proposals approved by the principal investigator.
Supporting Information: Study Protocol, ICF
Time Frame: Up to 3 years after manuscript publication
Access Criteria: Available to researchers with methodologically sound proposals approved by the principal investigator.

REFERENCES:
- [Derived] McCoy IE, Liu KD, Ghamarian E, Quenot JP, Zarbock A, Bihorac A, Khoo B, Gallagher MP, Du B, Joannidis M, Kashani K, Tolwani A, Bagshaw SM, Wald R; STandard versus Accelerated initiation of Renal Replacement Therapy in AKI (STARRT-AKI) Investigators. Dialysis Dependence in Standard versus Accelerated Initiation of KRT in AKI: A Post Hoc Analysis. Clin J Am Soc Nephrol. 2025 May 1;20(5):601-607. doi: 10.2215/CJN.0000000672. Epub 2025 Mar 11. PMID 40232884